CLINICAL TRIAL: NCT06988098
Title: Evaluation of the Effect of Different Deproteinizing Agents on the Clinical Success of Fissure Sealants in Permanent Teeth: Splint Mouth Clinical Study
Brief Title: The Effect of Different Deproteinising Agents on the Clinical Success of Fissure Sealants in Permanent Teeth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Alem Coşgun, Asistant proffessor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23-19
Record Dates: First submitted 2025-05-08; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Fissure Sealant
Keywords: Deproteinization Agents; Sodium Hypochlorite; Hypochlorous Acid; fissure sealent

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Hypochlorite, Wizard (Active Comparator): There are many studies in the literature showing that the use of 5.25% NaOCl as an enamel deproteinization agent is successful in positively affecting adhesion by removing organic elements from both the enamel structure and the pellicle on the enamel surface before acid application. However, sodium hypochlorite is a strong oxidizing agent and has disadvantages such as the risk of reaction in the soft tissues of the mouth, bad odor and bad taste, especially if not used carefully in pediatric dentistry, which has led to the search for an alternative material.
  Interventions: Other: application of deproteinization agents
- Hypochlorous Acid, Superox (Experimental): Hypochlorous acid is produced by the body's immune system cells, neutrophilic polymorphonuclear leukocytes, as a result of oxidative reactions to overcome pathogenic microorganisms and fight infection. Recently, slightly acidic HOCl solutions, developed by electrolysis of NaOCl, have been widely used as disinfectants. Hypochlorous acid has been shown to significantly reduce the lipopolysaccharide concentration of Porphyromonas gingivalis compared to NaOCl and chlorhexidine and to be an agent tolerated by oral tissues. It has also been reported that HOCl used as a mouthwash does not produce any systemic side effects. In clinical dentistry, HOCl has been shown to be highly effective as a result of its antimicrobial and deproteinizing properties. HOCl, with its low acidity, is an antiseptic irrigant with extraordinary properties, not only exhibiting biocompatibility and low cytotoxicity, but also having rapid and highly effective antimicrobial activity in physiological concentration rang
  Interventions: Other: application of deproteinization agents

INTERVENTIONS:
Other: application of deproteinization agents — Since there is no in vivo study in the literature evaluating the clinical success of the use of hypochlorous acid for deproteinization in fissure sealants, our planned study is the first in this regard.

SUMMARY:
Investigation of the effect of deproteinization agents on the clinical success of non-invasive fissure sealant application, which is a non-invasive method used to prevent caries formation or to stop the progression of initial caries lesions limited to enamel on tooth surfaces thought to be at high risk of caries.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 6-9 who do not have any systemic problems
* Have a score of 3 and 4 on the Frankl Behavior Scale
* Do not have a habit of clenching and/or grinding their teeth
* Have newly erupted permanent lower first molars without caries
* Have an indication for fissure sealant application

Exclusion Criteria:

* Teeth with fissure sealants
* Teeth with developmental defects such as hypoplasia
* Teeth with approximal or incipient caries lesions on one or both mandibular first permanent molars
* Children who are not systemically healthy
* Uncooperative children with scores of 1 and 2 on the Frankl Behavior Scale
* Children and parents who refuse to attend follow-up appointments
* Children with parafunctional habits such as teeth grinding

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Modified Simonsen Criteria | Following the sealant application, controls will be made at 6, 12, 24 and 36 months.
  Modified Simonsen Criteria
  Score 0 Fissure sealant is completely in the mouth and there is no new caries.
  Score 1 Partial loss of fissure sealant, no new caries.
  Score 2 Partial loss of fissure sealant and new caries.
  Score 3 Complete loss of fissure sealant, no new caries.
  Score 4 Complete loss of fissure sealant and new caries.

SECONDARY OUTCOMES:
Edge Integrity Evaluation Criteria | Following the sealant application, controls will be made at 6, 12, 24 and 36 months.
  Edge Integrity Evaluation Criteria
  0 The fissure sealant and tooth surface are intact and cannot be distinguished with a probe.
  1. The edges of the fissure sealants can be distinguished with a probe.
  2. There is a gap along the edge of the fissure sealant and deep cracks reaching the central fossa.

OTHER OUTCOMES:
Marginal Coloration Evaluation Criteria | Following the sealant application, checks will be made at 6, 12, 24 and 36 months
  Marginal Coloration Evaluation Criteria
  0 No color change between fissure sealant and tooth.
  1. Color change in only one area.
  2. Color change in many areas.
  3. Severe color change indicating leakage.
Anatomical Form Evaluation Criteria | Following the sealant application, checks will be made at 6, 12, 24 and 36 months
  Anatomical Form Evaluation Criteria
  0 Consistent with and continuous with occlusal form and structure.
  1. Change in anatomical form but all pits and fissures covered.
  2. a Partial loss of one or two pits or fissures but no need to repair or replace fissure sealant.
  2b Partial loss of pits and fissures, fissure sealant needs to be replaced or repaired.
  3 Loss of all pits and fissures.
  7 Partial loss due to occlusion
  9 Bleb not connected to margins

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpaşa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Feigal RJ, Musherure P, Gillespie B, Levy-Polack M, Quelhas I, Hebling J. Improved sealant retention with bonding agents: a clinical study of two-bottle and single-bottle systems. J Dent Res. 2000 Nov;79(11):1850-6. doi: 10.1177/00220345000790110601. PMID 11145354
- [Result] Simonsen RJ. Retention and effectiveness of dental sealant after 15 years. J Am Dent Assoc. 1991 Oct;122(10):34-42. doi: 10.14219/jada.archive.1991.0289. PMID 1835987

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT06988098/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT06988098/ICF_001.pdf